CLINICAL TRIAL: NCT04405518
Title: Impact of Two Thromboelastometry-guided Transfusion Strategies on Blood Product Requirements in Liver Transplantation. a Multicenter, Randomized Trial. TROMBOFIBtrial
Brief Title: Impact of Two Guided Transfusion Strategies on Blood Product Requirements in Liver Transplantation.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Antoni Sabaté Pes (Other)
Responsible Party: Sponsor-Investigator, Antoni Sabaté Pes, Head of Anesthesiology and Reanimation Department; MD; PhD, Hospital Universitari de Bellvitge
Organization: Hospital Universitari de Bellvitge (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TROMBOFIBtrial; 2018-002510-13 (EudraCT Number)
Record Dates: First submitted 2019-10-10; First posted 2020-05-28 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Fibrin Blood Clot
Keywords: fibrinogen; red blood cell pack transfusion; orthotopic liver transplantation
MeSH Terms: interventions — Fibrinogen

STUDY DESIGN:
Intervention Model Description: Participants will be randomly divided into a group receiving concentrate of fibrinogen in the different phases of the liver transplant procedure, to achieve
  * Thromboelastometry value (A10 FIBTEM) of 11mm (study group) or
  * Thromboelastometry value (A10 FIBTEM) of 8mm (control group) The doses of fibrinogen will be calculated acording to the formula based on previous study (AJT2017), rounded to the higher value according to the presentation format of the drug. Study medication will be stored at the hospital pharmacy.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Active Comparator): The doses of fibrinogen will be calculated acording to the formula based on previous study (AJT2017), rounded to the higher value according to the presentation format of the drug. Study medication will be stored at the hospital pharmacy.
  Formula: 8mm - A10FIBTEM registered in mm) x 1.1 = fibrinogen dose required
  Interventions: Drug: Fibrinogen Concentrate (Human) 1 MG [RiaSTAP]
- intervention group (Experimental): The doses of fibrinogen will be calculated acording to the formula based on previous study (AJT2017), rounded to the higher value according to the presentation format of the drug. Study medication will be stored at the hospital pharmacy.
  Formula: 11mm - A10FIBTEM registered in mm) x 1.1 = fibrinogen dose required
  Interventions: Drug: Fibrinogen Concentrate (Human) 1 MG [RiaSTAP]

INTERVENTIONS:
Drug: Fibrinogen Concentrate (Human) 1 MG [RiaSTAP] — The drug used in this study is Riastap, 1g (Fibrinogen). The dose administered will depend on the arm group assigned and in the results of the thromboelastogram during the procedure.

SUMMARY:
It is a national multicentre clinical study, where 3 hospitals are involved: Bellvitge University Hospital, Clinic Hospital of Barcelona and Cruces Hospital of Bilbao). It is a randomized study based on the Hemoglobin value of the patient with a 1:1 ratio, parallel groups, controlled and single blind, in patients undergoing an orthotopic liver transplant, confirming previously that the participants fulfill all the inclusion criteria and none of exclusion.

DETAILED DESCRIPTION:
A total of 176 patients will be included (88 per group) and each center can not include more than 40% of the sample to avoid bias.

Blood samples will be analyzed at different times of the surgical intervention by an electronic device called thromboelastogram. It evaluates the blood clot characteristics and, depending on the results, assesses the need to correct values by the administration of fibrinogen or platelets.

One of the coagulation parameter evaluated and corrected by thromboelastogram is called A10FIBTEM. In a previous study, the investigators have seen that maintaining some specific ranges in the A10FIBTEM, results in a decrease of the use of blood products. That's why the investigators have created 2 groups:

* The control group will be corrected up to a value of A10FIBTEM = 8mm.
* The intervention group will be corrected up to a value of A10FIBTEM = 11mm.

Subsequently, results between groups will be compared. The investigators have to consider that the drug used in this study (Riastap) is an authorized and commercial drug.

The main objective is to demonstrate that the administration of fibrinogen in the intervention group compared to the control group changes the administration of red blood cells pack during the liver transplant and in the first 24 hours after.

Secondary objectives consist in demonstrate that in the intervention group, there is also a change in the administration of other blood products, a change in acute renal damage, a change in hours of mechanical ventilation, no changes in thrombotic events in the hepatic graft or in the patient in the first 90 days of the liver transplant and no changes in re operations, re-transplantation, or mortality during the first 90 days of the liver transplant, compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Candidate to an orthotopic liver trasnplantation.
* Informed consent.
* Preoperative hemoglobine </= 130 g/L

Exclusion Criteria:

* Preoperative hemoglobin> 130 g / L
* Familial amyloid polyneuropathy
* Polycystosis hepatic
* Living donor liver transplant
* Uncontrolled donor after cardiac death
* Acute / subacute liver failure
* Re-transplant (in the same hospital admission)
* Use of Anticoagulation drugs before transplantation.
* Age <18 years.
* Pregnancy and lactation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2021-11-02 (Actual); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the rate of red blood cell packs transfusion during procedure and in the first 24hours after between groups. | Intraoperative and the first 24 hours after surgery.
  Demonstrate that the A10FIBTEM correction with the administration of fibrinogen up to an A10FIBTEM value of 11mm, change the administration of red blood cell pack during the procedure and in the first 24 hours after it, comparing to the administration of fibrinogen up to an A10FIBTEM of 8mm.

SECONDARY OUTCOMES:
Evaluation of the rate of other blood products between groups. | Intraoperative and the first 24 hours after surgery.
  Demonstrate that the A10FIBTEM correction with the administration of fibrinogen up to an A10 FIBTEM value of 11mm change the administration of platelets, frozen fresh plasma and other blood products.
Evaluation of the acute kidney injury between groups using the Kidney Disease Improving Global Outcomes scale,the minimum values is 1 and the maximum values is 3, higher scores mean a worse outcome. | first week after the procedure and until 90 days after the procedure.
  Demonstrate that the A10FIBTEM correction with the administration of fibrinogen up to an A10 FIBTEM value of 11mm change the kidney injury through study completion
Evaluation of the duration of mechanical ventilation in hours between groups. | first week after the procedure and until 90 days after the procedure..
  Demonstrate that the A10FIBTEM correction with the administration of fibrinogen up to an A10 FIBTEM value of 11mm change the need of mechanical ventilation through study completion (comparing the number of hours of mechanical ventilation of each group).
Number of participants with major advers cardiac events (MACE), Number of participants with, any sign of infection, Number of participants with neurological events through study completion | Until 90 days after the procedure.
  Demonstrate that the A10FIBTEM correction with the administration of fibrinogen up to an A10 FIBTEM value of 11mm change the Number of participants with any adverse events.
Number of participants with thrombotic events in the hepatic graft measured by ecodoppler assessment; and the number of participants with any other thrombotic events measured by ecodoppler assessment of leg extremity or tomography axial of the lungs | Until 90 days after procedure
  Demonstrate that the A10FIBTEM correction with the administration of fibrinogen up to an A10 FIBTEM value of 11mm do not change thrombotic events in the hepatic graft or in the patient.
Number of participants who require reoperation for any cause; Number of participants who require being re transplanted and number of participant who died through the study completion | Until 90 days after procedure
  Demonstrate that the A10FIBTEM correction with the administration of fibrinogen up to an A10 FIBTEM value of 11mm do not change the outcome related to reoperation, re-transplantations or mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Marta Caballero, Principal Investigator — Bellvitge University Hospital; Josep Beltran, Principal Investigator — Clinic Hospital, Barcelona; Rosa Gutierrez, Principal Investigator — Cruces Hospital, Bilbao
Locations (3):
- Spain (3):
  - Bellvitge Universitary Hospital, L'Hospitalet de Llobregat, Barcelone
  - Cruces Hospital, Bilbao, Vizcaya
  - Clinic Hospital, Barcelona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sabate A, Caballero M, Gutierrez R, Perez L, Vidal J, Llaurado S, Hereu P, Penafiel J, Blasi A. Factors associated with major complications defined by Clavien-Dindo classification 3-5 after liver transplantation: a prospective multicenter cohort study. Front Surg. 2025 Nov 14;12:1648512. doi: 10.3389/fsurg.2025.1648512. eCollection 2025. PMID 41321850